CLINICAL TRIAL: NCT03700866
Title: Evaluation of Functional Versus IADT Splinting Times on Tooth Mobility After Surgical Extrusion of Permanent Anterior Teeth: A Randomized Controlled Trial
Brief Title: Evaluation of Functional Versus IADT Splinting Times on Tooth Mobility After Surgical Extrusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maii Mohamed Mohamed Mohamed Ali, Assistant Lecturer of Pediatric Dentistry and Community Dentistry, Faculty of Dentistry, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: splinting time
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Dental Trauma
Keywords: luxation injury; splinting time; crown-root fracture; surgical extrusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Functional splinting time) (Experimental): Teeth with crown root fracture will be surgically extruded and splinted then the Periotest values will determine when the splint should be removed which will indicate the functional periodontal healing and as well the functional splinting time.
  The Periotest readings will be repeated with one week time interval between each series When the Periotest values of the traumatized tooth reach or even approximate the values of the corresponding normal tooth the splint will be removed.
  Interventions: Procedure: Functional splinting time
- (IADT splinting time) (Active Comparator): Teeth with crown root fracture in this group will be surgically extruded and splinted for two weeks according to the international association of dental traumatology (IADT) splinting time two ,weeks splinting, regardless the Periotest score.
  Interventions: Procedure: Functional splinting time

INTERVENTIONS:
Procedure: Functional splinting time — Functional splinting time is the time needed for the final healing and organization of Peridontal ligament of tooth with extrusive luxation injury to reattach to the alveolus and function normally in the oral cavity

SUMMARY:
The objective of this study is to compare functional splinting time effect versus the suggested splinting time of (IADT) effect on tooth mobility and possible healing outcomes for surgically extruded permanent anterior teeth with crown root fracture.

DETAILED DESCRIPTION:
Trauma involving the tooth supporting tissue, especially luxation injuries, is considered the most severe with consequences such as neurovascular disruption, pulp necrosis, and root resorption. Healing depends on factors such as the level of root development, the extent of damage to periodontal tissues, and the effects of bacterial contamination from the oral cavity .

The course of healing of the severed periodontal ligament will determine the treatment outcome of these injured teeth .As a result, all treatment procedures are directed to minimize undesired consequences which might lead not only to loss of tooth, but also to loss of alveolar bone.

The common treatment of luxated teeth is repositioning and splinting to achieve stability and to prevent further damage to the pulp and periodontal structures during healing. Splints should ensure adequate ﬁxation, prevent accidental ingestion or inhalation, and should protect teeth against traumatic forces during the vulnerable healing period .

The current guidelines for treatment of traumatic injuries by the International Association of Dental Traumatology (IADT) specify a short term functional splint for luxated teeth. However these protocols are based on clinical studies and animal experimentation employed rigid ﬁxation techniques so the results of these investigations are not representative of the current protocols . Also splinting times in IADT guidelines are derived mainly from animal studies which considered of low quality evidence .

As a result of, surgical tooth extrusion as treatment modality in cases of crown root fracture was chosen as a controlled traumatic injury to examine the true cause-effect relationship between splinting time and healing outcomes of periodontal ligament aiming to decrease the effect of bias, con-founders and probability of chance associated with the other types of luxation injury.

ELIGIBILITY:
Inclusion Criteria:

* Permanent anterior tooth/teeth with crown root fracture that needs surgical extrusion.
* Complicated or uncomplicated crown root fracture.
* Vital or necrotic tooth/ teeth.
* Mature or immature tooth /teeth.

Exclusion Criteria:

* Medically compromised patient
* Tooth suffered any type of luxation injury to decrease the risk of root resorption
* When root resorption is evident during the initial radiographic examination.
* Teeth with dilacerated root to avoid pulp necrosis and periapical infection that occur without any evident decay in these teeth as the central lumen of the root constitutes a pathway for bacteria.
* When root resorption is evident during the initial radiographic examination.
* Teeth with dilacerated root to avoid pulp necrosis and periapical infection that occur without any evident decay in these teeth as the central lumen of the root constitutes a pathway for bacteria.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-01-30 (Estimated); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
Tooth mobility | 3 months
  Tooth mobility will be assessed using Periotest the measurement unite is discrete range (-8 to 50)
Tooth mobility | 6 months
  Tooth mobility will be assessed using Periotest the measurement unite is discrete range (-8 to 50)
Tooth mobility | 9 months
  Tooth mobility will be assessed using Periotest the measurement unite is discrete range (-8 to 50)

SECONDARY OUTCOMES:
Root resorption | 9 months
  Root resorption will be assessed using digital radiography the outcome will be binary outcome (Present or Absent) using DIGORA software.
marginal bone resorption | 9 months
  marginal bone resorption will be assessed using digital radiography the outcome will be binary outcome (Present or Absent) using DIGORA software.